CLINICAL TRIAL: NCT05741866
Title: Protect PIVCs: An Adaptive Randomized Controlled Trial of a Novel Antimicrobial Dressing in Peripheral Intravenous Catheters (PIVCs).
Brief Title: Novel Antimicrobial Dressing in Peripheral Intravenous Catheters (PIVCs)
Acronym: ProP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Queensland (Other)
Collaborators: Queensland Children's Hospital (Other Government); Royal Brisbane and Women's Hospital (Other Government); University Hospital of Poitiers (Unknown); Griffith University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022/HE001952
Record Dates: First submitted 2022-12-15; First posted 2023-02-23 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2022-11

CONDITIONS: Vascular Access Complication; Device Related Infection; Device Related Sepsis; Device Site Reactions; Catheter Infection; Catheter Complications; Catheter-Related Infections; Catheter Related Complication; Occlusive Dressings; Wound Infection; Wound of Skin; Wound
Keywords: Peripheral Intravenous Catheter; PIVC; Intravenous; Vascular access device; randomised controlled trial; phlebitis; chlorhexidine gluconate; CHG dressing
MeSH Terms: conditions — Prosthesis-Related Infections; Catheter-Related Infections; Wound Infection; Wounds and Injuries; Phlebitis

STUDY DESIGN:
Intervention Model Description: A multi-centre, two-arm, parallel group adaptive randomised controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the intervention, blinding of patients/clinicians to the intervention is not possible. However, the statistician will be blinded for analysis; and the microbiologist and laboratory staff will also be blinded to treatment allocation when apportioning infection outcomes.
  Additionally, at the completion of Phase 1 (n=300) an independent data safety monitoring committee (DSMC) comprised of a biostatistician, physician and expert trialist, will review pre-defined blinded analyses, conducting a review of feasibility and safety data to determine if the trial should continue to a fully powered RCT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control (Active Comparator): Bordered Polyurethane Dressing
  Interventions: Device: Standard bordered polyurethane dressing
- Intervention (Experimental): CHG Bordered Polyurethane Dressing
  Interventions: Device: Chlorhexidine gluconate impregnated bordered polyurethane dressing

INTERVENTIONS:
Device: Chlorhexidine gluconate impregnated bordered polyurethane dressing — PIVCs will be dressed and secured at the participating sites
  * RBWH and PUH: PIVCs will be dressed with Tegaderm™ Antimicrobial I.V. Advanced Securement (9132) dressing and secured with non-sterile tape over extension tubing.
  * QCH: PIVCs will be dressed with Tegaderm™ Antimicrobial I.V. Advanced Securement (9132) dressing and secured with tubular bandage +/- arm board and non-sterile stretchy tape if PIVC over flexible joint, +/- tissue adhesive as per clinician preference.
  Other Names: Tegaderm™ Antimicrobial I.V. Advanced Securement (9132)
  Arms: Intervention
Device: Standard bordered polyurethane dressing — PIVCs will be dressed and secured as per standard practice at the participating sites
  * RBWH and PUH: Bordered polyurethane dressing (Tegaderm™ IV Advanced 1683) and non-sterile tape strip over extension tubing.
  * QCH: Bordered polyurethane dressing (Tegaderm™ IV Advanced 1682 or 1683) and secured with tubular bandage +/- arm board and non-sterile stretchy tape if PIVC over flexible joint, +/- tissue adhesive as per clinician preference.
  Other Names: Tegaderm™ IV Advanced (1682 or 1683)
  Arms: Control

SUMMARY:
The goal of this clinical trial is to compare a chlorhexidine impregnated dressing for peripheral intravenous catheters (PIVCs) to the standard dressing currently used in general medical and surgical inpatient wards.

The main questions it aims to answer are:

* Study Feasibility
* Occurrence of infectious complications related to the PIVC

Participants will be randomly allocated to receive either of the below dressings to cover and secure their PIVC:

* The standard dressing used at their hospital, or
* The intervention dressing which has Chlorhexidine gluconate (CHG) on it

Researchers will compare standard and CHG dressings to see if the presence of CHG improves the occurrence of infectious complications related to the PIVC.

DETAILED DESCRIPTION:
This study is a multi-centre, two-arm, parallel group adaptive Randomized Controlled Trial (RCT) to test effectiveness, cost-effectiveness, and safety of 3M™ Tegaderm™ Antimicrobial IV Advanced Securement dressings with standard polyurethane dressings for PIVCs. The study has two phases. Phase I is an internal feasibility pilot for which only feasibility outcomes will be considered (no analysis). At this time (n=300) an independent Data Safety Monitoring Committee (DSMC) comprised of a biostatistician, physician and expert trialist will review pre-defined blinded analyses of feasibility and safety data. Phase II will then go ahead if feasibility outcomes are satisfactory, and will involve continuation of trial recruitment to complete a definitive RCT. If Phase II does not proceed then all outcomes will be reported at the end of Phase I.

Setting and sample:

Australia: The ProP Trial will be undertaken in the general medical/surgical and oncology/hematology departments at the Queensland Children's Hospital (QCH; Site 1), and the general medical/surgical departments at the Royal Brisbane and Women's Hospital (RBWH; Site 2) Brisbane, Australia. These are both large quaternary referral teaching hospitals (Site 1: 359 beds; Site 2: 929 beds).

France: The ProP Trial will be undertaken in the University Hospital of Poitiers (PUH), a large referral teaching hospital with 959 acute beds. Patients will be recruited at the Emergency Department, before being admitted to medical wards.

Sample size:

Phase 1: The investigators will recruit 300 patients (200 Australia and 100 France) with 150 patients per arm. This sample size is not determined by statistical power but to test protocol feasibility and gain estimates of effect to inform a sample size calculation for a full trial. The investigators aim to recruit 300 patients over 16 weeks (19 per week).

Phase 2: The investigators will continue recruitment to the sample size recommended by the DSMC and the Trial Steering Committee. The investigators anticipate this will be no more than a sample of 2624 patients (1312/group) which would have 90% power to detect an absolute 5% reduction in the primary outcome from 22% to 17% (2-way alpha 0.05) (http://powerandsamplesize.com/calculators).

ELIGIBILITY:
Inclusion Criteria:

* PIVC to be inserted with expected dwell >48 hours
* Provided written and informed consent (patient or carer)

Australia only

• ≥6 years of age (due to size of dressing)

France only

• ≥18 years of age

Exclusion Criteria:

* Burned, non-intact or scarred skin at the insertion site
* Known allergy to CHG or transparent dressing adhesives
* Palliative care patients on end-of-life pathway
* Patient who has already participated in the study
* Placement of a PIVC in an emergency, that does not allow the usual rules of hygiene for insertion to be adhered to.

Additional exclusions to Australian study only

* Non-English-speaking patients without interpreter
* Under the care of Child and Family Services and unable to gain consent from case worker (paediatric patients)

Additional exclusions to French study only

* Patients not benefiting from the French Social Security scheme or not benefiting from it through a third party,
* Persons benefiting from enhanced protection, namely minors, persons deprived of their liberty by a judicial or administrative decision, adults under legal protection.
* Known pregnant or breastfeeding women
* Predictably difficult vascular access (IV drug addiction, obesity)

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility for a definitive RCT | On completion of 300 participants
  The feasibility of conducting a definitive RCT will be assessed against the following criteria:
  i. Study Eligibility as per inclusion/exclusion criteria (≥80% of screened participants will be eligible for study inclusion) ii. Participant Recruitment onto study (≥80% of eligible participants will provide informed consent to participate in the study) iii. Retention of study participants (<10% will be lost to follow up) iv. Protocol fidelity of study participants (≥80% will receive the allocated intervention) v. Missing data for primary outcome 2 (<5% of primary outcome 2 data will be unable to be collected) vi. Satisfaction of participants/parents and staff (<10% report "low" satisfaction with the intervention arm (rated low/medium/high) vii. An estimate of catheter-related infectious complications (defined as per primary outcome 2) in the control group that indicate a fully powered multi-site RCT is achievable
Catheter-related infectious complications and phlebitis | Daily until 48hours after study PIVC is removed.
  Proportion of patients with a composite measure of PIVC Colonization; PIVC local infection; PIVC-associated Bloodstream Infection (BSI) and Phlebitis. These measures are defined below in secondary outcomes.
  If patients meet more than one of the following [e.g., phlebitis and PIVC local infection], both will be collected however only counted once for the composite measure.

SECONDARY OUTCOMES:
PIVC tip colonization | Daily until 48hours after study PIVC is removed.
  >15 cfu of a pathogen semi-quantitative method, or ≥1000 cfu of a pathogen per mL broth method.
  PIVC tips will be collected based on Nurse and laboratory availability at time of PIVC removal.
PIVC local infection without Bloodstream Infection (BSI) | Daily until 48hours after study PIVC is removed.
  Proportion of patients with a PIVC local infection without BSI as defined by NHSN 2021 criteria for Cardiovascular System VASC-Arterial or Venous Infection (CVS-VASC); adult and child/infant criteria.
  Collected daily by either the research nurse or medical investigators from either direct observation, consultation with the clinical staff or review of the medical record and microbiology results.
PIVC-associated Bloodstream Infection | Daily until 48hours after study PIVC is removed.
  Proportion of patients with a laboratory Confirmed Bloodstream Infection, as defined by NHSN 2021 adult and infant criteria
  Collected daily by either research nurse or medical investigators from either direct observation, consultation with the clinical staff or review of the medical record and microbiology results.
Phlebitis | Daily until 48hours after study PIVC is removed.
  Either pain or tenderness [>1 on a scale of 0 to 10]), or at least 2 of erythema, swelling, purulence or palpable cord.
  Collected daily by either research nurse or medical investigators from either direct observation, consultation with the clinical staff or review of the medical record.
PIVC device failure | Daily until 48hours after study PIVC is removed.
  Proportion of patients, a composite of infiltration/ extravasation, blockage/occlusion (with/without leakage), phlebitis (as defined above), thrombosis, dislodgement (complete/partial) or infection (as defined above).
  Collected daily by either research nurse or medical investigators from either direct observation, consultation with the clinical staff or review of the medical record.
Dressing durability | Daily until study PIVC is removed.
  Proportion of patients with dressing durability assessed as:
  (i) the dressing remains adhered to the skin on all four sides until PIVC removal; and, (ii) accidental dislodgement (excluding patients who deliberately remove their PIVC).
  Collected daily by either research nurse or medical investigators from either direct observation, consultation with the clinical staff or review of the medical record.
Skin colonization | On study PIVC removal
  Reported semi-quantitatively as scant, 1+, 2+, 3.
  PIVC skin swabs will be collected based on Nurse and laboratory availability at time of PIVC removal.
Adverse skin event | Daily until 48hours after study PIVC is removed.
  Proportion of patients with skin complications at PIVC site: mechanical (e.g. pressure injury, skin tears, blisters, bruising) or inflammatory complications (e.g. contact/allergic dermatitis, skin rash, pruritus).
  Collected daily by either research nurse or medical investigators from either direct observation, consultation with the clinical staff or review of the medical record.
Serious adverse event | Daily until 48hours after study PIVC is removed.
  Proportion of patients with anaphylactic reaction to CHG in dressing; or mortality related to PIVC infection.
  Collected daily by either research nurse or medical investigators from either direct observation, consultation with the clinical staff or review of the medical record.
Cost effectiveness | Until discharge.
  Direct and indirect healthcare costs to the health system, including cost per complication avoided.
  Collected daily by either research nurse or medical investigators from either direct observation, consultation with the clinical staff or review of the medical record and microbiology results.
  A random subset of 15% of participants will have all subsequent devices recorded until completion of treatment for the participant's current admission. Date of discharge will be recorded for all participants to calculate length of stay.
Patient reported experience measures of the dressing | Daily until 48hours after study PIVC is removed.
  Proportion of participants/parents who report their satisfaction with the dressing rated low/medium/high with respective prompts of:
  1. "I'd rather use a different dressing next time"
  2. "The dressing was ok, but I'm happy to try other types"
  3. "It was a really good dressing and I'd like to use this one again"
  A Patient-Reported Experience Measure survey will be conducted on study PIVC removal.
  Patient's will have the opportunity to comment on the dressing and their satisfaction with it at any time during study participation.
Clinician reported experience measures of the dressing including application and removal | Daily until 48hours after study PIVC is removed.
  Proportion of clinicians who report their satisfaction with the dressing rated low/medium/high with respective prompts of:
  1. "I'd rather use a different dressing next time"
  2. "The dressing was ok, but I'm happy to try other types"
  3. "It was a really good dressing and I'd like to use this one again"
  Collected opportunistically between dressing application to 48 hours after study PIVC removal.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Rickard, Principal Investigator — The University of Queensland
Locations (3):
- Australia (2):
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Queensland Children's Hospital, South Brisbane, Queensland
- University Hospital of Poitiers, Poitiers, Nouvelle-Aquitaine, France

IPD SHARING:
Plan to Share IPD: Yes
Available to individuals who provide a methodologically sound proposal and at the discretion of the Principal Investigator.

REFERENCES:
- [Derived] Rickard CM, Drugeon B, Ullman A, Marsh NM, Corley A, Ball D, O'Brien C, Kleidon TM, Guenezan J, Couvreur R, McCarthy KL, Seguin S, Batiot G, Byrnes J, Schults J, Zahir SF, Mimoz O. Protect peripheral intravenous catheters: a study protocol for a randomised controlled trial of a novel antimicrobial dressing for peripheral intravenous catheters (ProP trial). BMJ Open. 2024 Jul 16;14(7):e084313. doi: 10.1136/bmjopen-2024-084313. PMID 39013653